CLINICAL TRIAL: NCT00776919
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Active And Vehicle-Controlled Study Of The Safety And Efficacy Of A Clindamycin / Benzoyl Peroxide Gel Versus Clindamycin Gel Versus Benzoyl Peroxide Gel Versus Vehicle Gel In Subjects With Acne Vulgaris
Brief Title: Trial of Clindamycin / Benzoyl Peroxide Gel in Subjects With Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: Rho, Inc. (Industry); Quintiles, Inc. (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114677
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): clindamycin / benzoyl peroxide gel
  Interventions: Drug: clindamycin / benzoyl peroxide gel
- 2 (Active Comparator): Clindamycin gel
  Interventions: Drug: clindamycin gel
- 3 (Active Comparator): BPO gel
  Interventions: Drug: BPO gel
- 4 (Placebo Comparator): vehicle gel
  Interventions: Drug: vehicle gel

INTERVENTIONS:
Drug: clindamycin / benzoyl peroxide gel — Once a day application to the face
  Arms: 1
Drug: clindamycin gel — Once a day application to the face
  Arms: 2
Drug: BPO gel — Once a day application to the face
  Arms: 3
Drug: vehicle gel — Once a day application to the face
  Arms: 4

SUMMARY:
This is a Randomized, Double-Blind, Controlled Study to evaluate the Safety and Efficacy of a clindamycin / benzoyl peroxide gel in Subjects with Acne Vulgaris

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, comparator and vehicle-controlled study in subjects with acne vulgaris. Approximately 1320 subjects will be enrolled. Subjects will be randomized to 1 of 4 parallel study groups in a 1:1:1:1 ratio (clindamycin / benzoyl peroxide gel:clindamycin gel:BPO gel:vehicle gel).

ELIGIBILITY:
Inclusion Criteria:

* Be 12 to 45 years of age, inclusive, and in good general health.
* Clinical diagnosis of acne vulgaris
* Females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product.
* Have the ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study.
* Have the ability to understand and sign a written informed consent form, which must be completed prior to study specific tasks being performed. Subjects under the legal age of consent in the state/province/country where the study is conducted must provide assent and have the written informed consent of a parent or guardian.

Exclusion Criteria:

* Are pregnant or breast-feeding.
* Have a history or presence of other conditions that may increase the risk of the subject participating in the study and/or affect the evaluated outcomes.
* Used topical antibiotics on the face or used systemic antibiotics within the past 2 weeks.
* Used topical corticosteroids on the face or systemic corticosteroids within the past 4 weeks. Use of inhaled, intra-articular, or intra-lesional steroids other than for facial acne is acceptable.
* Used systemic retinoids within the past 6 months or topical retinoids within the past 6 weeks.
* Received treatment with estrogens (including oral, implanted, injected and topical contraceptives), androgens, or anti-androgenic agents for 12 weeks or less immediately prior to starting study product. Subjects who have been treated with estrogens, as described above, androgens, or anti-androgenic agents for more than 12 consecutive weeks prior to start of study product are allowed to enroll as long as they do not expect to change dose, drug, or discontinue use during the study.
* Used topical anti-acne medications (eg, BPO, azelaic acid, resorcinol, salicylates, etc.) within the past 2 weeks.
* Used abradents or facial procedures, within the past 2 weeks.
* Use medications that may exacerbate acne.
* Have a known hypersensitivity or have had previous allergic reaction to any of the active components, lincomycin, or excipients of the study product.
* Used any investigational therapy within the past 4 weeks, or currently participating in another clinical study.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1315 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (16):
  - Rady Children's Hospital San Diego, Div. of Pediatric & Adolescents Dermatology, San Diego, California
  - The Laser Institute for Dermatology, Santa Monica, California
  - Cherry Creek Research, Inc., Denver, Colorado
  - Skin Care Research, Inc., Boca Raton, Florida
  - FXM Research, Miami, Florida
  - University of Miami Cosmetic Medicine and Research Institute, Miami Beach, Florida
  - Atlanta Dermatology & Vein Research Center, LLC, Alpharetta, Georgia
  - SKINQRI, Lincolnshire, Illinois
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - DermResearch, PLLC, Louisville, Kentucky
  - Somerset Skin Centre, Troy, Michigan
  - Dermatology Associates of Rochester, PC, Rochester, New York
  - DermResearch Center of New York, Stony Brook, New York
  - The Skin Wellness Center, PC, Knoxville, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - Progressive Clinical Research, San Antonio, Texas
- Belize (2):
  - Dermatology and Skin Care Center FXM Research International, Belize City
  - Dr. Moguel's Clinic/FXM Research International, Belize City
- Canada (6):
  - Guildford Dermatology Specialist, Surrey, British Columbia
  - Dermatrial Research, Hamilton, Ontario
  - Lynderm Research, Inc., Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - CRDQ Centre de Recherche Dermatologique du Quebec, Québec, Quebec
  - Nexus Clinical Research, St. John's

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Eichenfield LF, Alio Saenz AB. Safety and efficacy of clindamycin phosphate 1.2%-benzoyl peroxide 3% fixed-dose combination gel for the treatment of acne vulgaris: a phase 3, multicenter, randomized, double-blind, active- and vehicle-controlled study. J Drugs Dermatol. 2011 Dec;10(12):1382-96. PMID 22134562
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 114677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Duac Low-dose (LD) Gel: Duac LD gel (combination of 1% clindamycin phosphate and 3% benzoyl peroxide) applied once daily (in the morning or evening, but at approximately the same time each day) to the entire face for 12 weeks
- Clindamycin Gel: Clindamycin gel (containing 1% clindamycin phosphate) applied once daily (in the morning or evening, but at approximately the same time each day) to the entire face for 12 weeks
- BPO Gel: Benzoyl peroxide (BPO) gel (containing 3% benzoyl peroxide) applied once daily (in the morning or evening, but at approximately the same time each day) to the entire face for 12 weeks
- Vehicle Gel: Matching vehicle gel without the active ingredients clinidamycin phosphate and benzoyl peroxide, applied once daily (in the morning or evening, but at approximately the same time each day) to the entire face for 12 weeks
Period: Overall Study
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Started | 327 | 328 | 328 | 332
Completed | 300 | 295 | 296 | 293
Not Completed | 27 | 33 | 32 | 39
Not completed — Withdrawal by Subject | 16 | 14 | 15 | 26
Not completed — Lost to Follow-up | 8 | 12 | 11 | 8
Not completed — Adverse Event | 1 | 0 | 2 | 2
Not completed — Protocol Violation | 1 | 2 | 0 | 1
Not completed — Other: Lack of Efficacy/Lost Medication | 1 | 5 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel | Total
Number analyzed (Participants) | 327 | 328 | 328 | 332 | 1315
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.0 (7.0) | 20.2 (6.9) | 20.6 (7.1) | 20.7 (7.4) | 20.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 180 | 203 | 210 | 795
  Male | 125 | 148 | 125 | 122 | 520
Race/Ethnicity, Customized [Number; unit: participants]
  White | 259 | 274 | 251 | 258 | 1042
  Black | 47 | 37 | 54 | 54 | 192
  Asian | 13 | 9 | 17 | 16 | 55
  Multiracial | 5 | 7 | 7 | 4 | 23
  American Indian or Alaska Native | 3 | 1 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement of at Least 2 Grades in the Investigator's Static Global Assessment (ISGA) Score From Baseline to Week 12
Description: During each study visit, investigators/assessors evaluated acne severity of the participants' faces using the ISGA scale: 0=clear skin with no lesions (L); 1=almost clear, rare non-inflammatory L; 2=mild, some non-inflammatory L with no more than a few inflammatory L, no nodular L; 3=moderate, many non-inflammatory L, may have some inflammatory L, but no more than 1 small nodular L; 4=severe, many non-inflammatory and inflammatory L, but no more than a few nodular L; 5=very severe, many non-inflammatory and inflammatory L, and more than a few nodular L.
Time Frame: Baseline (Day 1) and Week 12
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to and received at least 1 application of study product. Participants with missing Week 12 evaluations were considered failures. Failures are defined as those participants with a 1-grade improvement, no improvement, or a worsening.
Measure: Number; unit: participants
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 327 | 328 | 328 | 332
participants | 129 | 82 | 100 | 59
Statistical Analysis 1: Comparison: Duac Low-dose (LD) Gel vs Clindamycin Gel; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Duac Low-dose (LD) Gel vs BPO Gel; Test type: Superiority or Other; p = 0.016, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Duac Low-dose (LD) Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Primary Outcome: Mean Change From Baseline (BL) to Week 12 in Inflammatory Lesion Counts
Description: During each study visit, trained study personnel at every investigational center assessed the inflammatory (pustules [small inflamed elevation of the skin that is filled with pus], papules [solid elevation of skin with no visible fluid], nodules [larger than papules with significant depth]) lesion counts for each participant. Each type of lesion was counted separately, and counts were taken from the face (including forehead, nose, cheeks, and chin). Missing values were imputed using the last observation carried forward (LOCF) method.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT Population. Participants who missed >=16 days of treatment or reported lost medication and never began treatment were excluded from the analysis. In the LOCF method, the last available observation, including BL, was used to estimate subsequent missing data points.
Measure: Mean (Standard Deviation); unit: lesion counts
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 322 | 318 | 323 | 329
lesion counts | -18.2 (10.4) | -15.6 (11.6) | -16.8 (11.5) | -13.1 (12.1)
Statistical Analysis 1: Comparison: Duac Low-dose (LD) Gel vs Clindamycin Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — Based on an analysis of covariance (ANCOVA) with factors of treatment, center, and interaction of treatment-center. If the treatment-center interaction was not significant at the 0.1 level, this interaction was excluded from the ANCOVA model
Statistical Analysis 2: Comparison: Duac Low-dose (LD) Gel vs BPO Gel; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Duac Low-dose (LD) Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

3. Primary Outcome: Mean Change From Baseline to Week 12 in Non-inflammatory Lesion Counts
Description: During each study visit, trained study personnel at every investigational center assessed the non-inflammatory (open comedones [blackheads] and closed comedones [whiteheads]) lesion counts for each participant. Each type of lesion was counted separately, and counts were taken from the face (including forehead, nose, cheeks, and chin).
Time Frame: Baseline (Day 1) and Week 12
Population: ITT Population. Participants who missed >=16 days of treatment or who reported they had lost their medication and never began treatment were excluded from the analysis. Missing values for all other participants were imputed using the LOCF method.
Measure: Mean (Standard Deviation); unit: lesion counts
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 322 | 318 | 323 | 329
lesion counts | -24.8 (20.1) | -19.8 (19.8) | -22.2 (17.6) | -14.8 (21.6)
Statistical Analysis 1: Comparison: Duac Low-dose (LD) Gel vs Clindamycin Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Duac Low-dose (LD) Gel vs BPO Gel; Test type: Superiority or Other; p = 0.102, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Duac Low-dose (LD) Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

4. Primary Outcome: Mean Change From Baseline to Week 12 in Total Lesion Counts
Description: During each study visit, trained study personnel at every investigational center assessed the inflammatory (pustules, papules, nodules) and non-inflammatory (open and closed comedones) lesion counts for each participant. Each type of lesion was counted separately; the lesion counts were taken from the face (including forehead, nose, cheeks, and chin). Total lesion counts were calculated as the sum of the inflammatory and non-inflammatory lesion counts.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: lesion counts
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 322 | 318 | 323 | 329
lesion counts | -43.0 (27.1) | -35.5 (27.1) | -39.0 (25.0) | -27.8 (29.8)
Statistical Analysis 1: Comparison: Duac Low-dose (LD) Gel vs Clindamycin Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Duac Low-dose (LD) Gel vs BPO Gel; Test type: Superiority or Other; p = 0.032, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Duac Low-dose (LD) Gel vs Vehicle Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]

5. Secondary Outcome: Mean Percent Change From Baseline to Week 12 in Lesion Counts (Total, Inflammatory, and Non-inflammatory)
Description: During each study visit, trained study personnel at every investigational center assessed the inflammatory (pustules, papules, nodules) and non-inflammatory (open and closed comedones) lesion counts for each participant. Each type of lesion was counted separately; the lesion counts were taken from the face (including forehead, nose, cheeks, and chin). Total lesion counts were calculated as the sum of the inflammatory and non-inflammatory lesion counts. Percent change from Baseline to Week 12 was calculated as the value at Week 12 minus the value at Baseline divided by the Baseline value * 100.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change in lesion counts
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 322 | 318 | 323 | 329
Percent change in lesion counts
  Inflammatory Lesions | -68.9 (29.6) | -58.1 (35.8) | -61.8 (31.5) | -48.8 (37.1)
  Non-inflammatory Lesions | -53.9 (32.2) | -43.3 (39.6) | -50.8 (33.5) | -34.0 (47.2)
  Total Lesions | -59.8 (28.0) | -49.2 (33.8) | -55.5 (28.8) | -40.4 (37.5)

6. Secondary Outcome: Number of Participants Who Had a Subject Global Assessment (SGA) Score of 0 or 1 at Week 12
Description: During each study visit, participants evaluated their facial acne (excluding the scalp) using the SGA scale: 0=free of acne, with only an occasional blackhead/whitehead; 1=several blackheads/whiteheads and small pimples, no tender deep-seated bumps/cysts; 2=several to many blackheads/whiteheads and small to medium-sized pimples, one deep-seated bump/cyst; 3=many blackheads/whiteheads, many medium- to large-sized pimples, few deep-seated bumps/cysts; 4=presence of blackheads/whiteheads, several to many medium- to large-sized pimples, deep-seated bumps/cysts dominate.
Time Frame: Week 12
Population: ITT Population. Participants with missing Week 12 evaluations were considered failures. Failures were defined as those participants with an SGA score >=2.
Measure: Number; unit: participants
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 327 | 328 | 328 | 332
participants | 209 | 171 | 189 | 154

7. Secondary Outcome: Number of Participants Who Had an ISGA Score of 0 or 1 at Week 12
Description: During each study visit, investigators/assessors evaluated the acne severity of participants' faces using the ISGA scal: 0=clear skin with no lesions (L); 1=almost clear, rare non-inflammatory L; 2=mild, some non-inflammatory L with no more than a few inflammatory L, no nodular L; 3=moderate, many non-inflammatory L, may have some inflammatory L, but no more than 1 small nodular L; 4=severe, many non-inflammatory and inflammatory L, but no more than a few nodular L; 5=very severe, many non-inflammatory and inflammatory L, and more than a few nodular L.
Time Frame: Week 12
Population: ITT Population. Participants with missing Week 12 evaluations were considered failures. Failures were defined as those participants with an ISGA score >=2.
Measure: Number; unit: participants
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 327 | 328 | 328 | 332
participants | 148 | 91 | 116 | 81

8. Secondary Outcome: Mean Change From Baseline to Week 12 in Systolic and Diastolic Blood Pressure
Description: Systolic and diastolic blood pressure were measured at Baseline and Week 12 (end of study). Mean change from Baseline was calculated as the mean value at Week 12 minus the mean value at Baseline.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT Population. Only those participants with data available at both Baseline and Week 12 were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 305 | 302 | 305 | 309
Millimeters of mercury (mmHg)
  Systolic blood pressure | 0 (10) | 0 (11) | 0 (12) | 0 (10)
  Diastolic blood pressure | 0 (8) | 1 (9) | 0 (8) | 0 (8)

9. Secondary Outcome: Mean Change From Baseline to Week 12 in Temperature
Description: Temperature was measured at Baseline and Week 12 (end of study). Mean change from Baseline was calculated as the mean value at Week 12 minus the mean value at Baseline.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT Population. Only those participants with data available at both Baseline and Week 12 were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees centigrade
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 304 | 302 | 305 | 309
Degrees centigrade | -0.1 (0.4) | 0.0 (0.4) | 0.0 (0.4) | 0.0 (0.4)

10. Secondary Outcome: Mean Change From Baseline to Week 12 in Pulse Rate
Description: Pulse rate was measured at Baseline and Week 12 (end of study). Mean change from Baseline was calculated as the mean value at Week 12 minus the mean value at Baseline.
Time Frame: Baseline (Day 1) and Week 12
Population: ITT Population. Only those participants with data available at both Baseline and Week 12 were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 305 | 302 | 304 | 309
Beats per minute (bpm) | 1 (10) | 2 (11) | 2 (9) | 2 (11)

11. Secondary Outcome: Mean Change From Baseline to Weeks 2, 4, 8, and 12 in Erythema, Dryness, and Peeling
Description: Erythema (Er, redness), dryness (Dr), and peeling (Pn), were evaluated independently by the investigator as: 0 (absent)=no Er, Dr, or Pn; 1 (slight)=faint red/pink coloration (col.), barely perceptible Dr with no flakes or fissure, mild localized Pn; 2 (mild)=light red/pink col., perceptible Dr with no flakes/fissure, mild and diffuse Pn; 3 (moderate)=medium red col., easily noted Dr and flakes but no fissure; 4 (severe)=beet red col., Dr with flakes and fissure, prominent dense Pn. Change from Baseline was calculated as the value at Weeks 2, 4, 8, and 12 minus the the value at Baseline.
Time Frame: Baseline; Weeks 2, 4, 8, and 12
Population: ITT Population. Only those participants with data available at both Baseline and the indicated assessment week were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 298 | 302 | 306 | 306
scores on a scale
  Erythema, Week 2, n=298, 302, 306, 306 | -0.05 (0.63) | -0.01 (0.58) | -0.07 (0.56) | -0.02 (0.61)
  Erythema, Week 4, n=298, 300, 299, 306 | -0.07 (0.66) | -0.07 (0.64) | -0.08 (0.67) | -0.06 (0.64)
  Erythema, Week 8, n=297, 296, 294, 293 | -0.12 (0.71) | -0.08 (0.67) | -0.15 (0.68) | -0.08 (0.73)
  Erythema, Week 12, n=297, 296, 296, 294 | -0.17 (0.66) | -0.18 (0.63) | -0.17 (0.67) | -0.13 (0.69)
  Dryness, Week 2, n=298, 302, 306, 306 | 0.07 (0.54) | 0.03 (0.48) | 0.09 (0.61) | 0.04 (0.50)
  Dryness, Week 4, n=298, 300, 299, 306 | 0.05 (0.58) | -0.02 (0.51) | 0.08 (0.55) | 0.00 (0.52)
  Dryness, Week 8, n=297, 296, 294, 293 | 0.00 (0.53) | -0.02 (0.58) | 0.05 (0.57) | 0.02 (0.56)
  Dryness, Week 12, n=297, 296, 296, 294 | -0.07 (0.62) | -0.10 (0.53) | -0.01 (0.57) | -0.04 (0.55)
  Peeling, Week 2, n=298, 302, 306, 306 | 0.03 (0.43) | 0.02 (0.36) | 0.08 (0.51) | 0.02 (0.41)
  Peeling, Week 4, n=298, 300, 299, 306 | -0.01 (0.39) | 0.00 (0.36) | 0.01 (0.39) | 0.00 (0.40)
  Peeling, Week 8, n=297, 296, 294, 293 | -0.01 (0.41) | -0.01 (0.42) | -0.01 (0.40) | 0.00 (0.43)
  Peeling, Week 12, n=297, 296, 296, 294 | -0.08 (0.44) | -0.06 (0.40) | -0.02 (0.50) | -0.04 (0.43)

12. Secondary Outcome: Mean Change From Baseline to Weeks 2, 4, 8, and 12 in Itching and Burning/Stinging
Description: Itching and burning/stinging (piercing pain) were evaluated independently by the investigator as: 0 (none)=normal, no discomfort; 1 (slight)=noticeable discomfort that caused intermittent awareness; 2 (moderate)=noticeable discomfort that caused intermittent awareness and interfered occasionally with normal daily activities; 3 (strong)=definite continuous discomfort that interfered with normal daily activities. Change from Baseline was calculated as the value at Weeks 2, 4, 8, and 12 minus the value at Baseline.
Time Frame: Baseline; Weeks 2, 4, 8, and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 298 | 302 | 306 | 306
scores on a scale
  Itching, Week 2, n=297, 301, 305, 305 | -0.11 (0.67) | -0.18 (0.67) | -0.04 (0.64) | -0.06 (0.65)
  Itching, Week 4, n=298, 299, 299, 305 | -0.11 (0.67) | -0.18 (0.68) | -0.07 (0.68) | -0.10 (0.61)
  Itching, Week 8, n=297, 295, 293, 291 | -0.16 (0.75) | -0.24 (0.69) | -0.08 (0.68) | -0.08 (0.62)
  Itching, Week 12, n=297, 295, 294, 293 | -0.21 (0.70) | -0.28 (0.67) | -0.13 (0.72) | -0.13 (0.63)
  Burning/Stinging, Week 2, n=297, 301, 305, 305 | 0.02 (0.58) | -0.06 (0.48) | -0.02 (0.56) | -0.05 (0.53)
  Burning/Stinging, Week 4, n=298, 2991, 299, 305 | -0.06 (0.57) | -0.09 (0.46) | -0.05 (0.55) | -0.02 (0.59)
  Burning/Stinging, Week 8, n=297, 295, 293, 291 | -0.05 (0.57) | -0.09 (0.46) | -0.05 (0.55) | -0.06 (0.54)
  Burning/Stinging, Week 12, n=297, 295, 294, 293 | -0.09 (0.58) | -0.13 (0.48) | -0.04 (0.60) | -0.04 (0.49)

13. Secondary Outcome: Mean Duration of Study Product Use
Description: Mean duration of study product use was calculated as the average total duration inclusive of missed applications of the study product.
Time Frame: Baseline (Day 1) through Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 327 | 328 | 328 | 332
days | 79.5 (16.4) | 78.0 (17.9) | 78.0 (18.4) | 77.8 (18.4)

14. Secondary Outcome: Number of Participants Reporting the Indicated Treatment-emergent Adverse Events (AEs) Resulting in Study Product Discontinuation
Description: An AE included, but was not limited to, any clinically significant worsening of a pre-existing condition; an event occurring from overdose (i.e., a dose higher than that indicated in the protocol) of the study product, whether accidental or intentional; an event occurring from abuse (e.g., use for nonstudy reasons) of the study product; or an event that was associated with the discontinuation of the use of the study product.
Time Frame: Baseline (Day 1) through Week 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Number analyzed (Participants) | 327 | 328 | 328 | 332
participants
  Application Site Dermatitis | 1 | 0 | 0 | 0
  Application Site Hypersensitivity | 0 | 0 | 1 | 0
  Application Site Pruritus | 0 | 0 | 1 | 1
  Varicella | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Duac Low-dose (LD) Gel | Clindamycin Gel | BPO Gel | Vehicle Gel
Serious Adverse Events (participants affected / at risk) | 0/327 | 0/328 | 1/328 | 0/332
Other Adverse Events (participants affected / at risk) | 72/327 | 83/328 | 102/328 | 87/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duac Low-dose (LD) Gel (N=327) | Clindamycin Gel (N=328) | BPO Gel (N=328) | Vehicle Gel (N=332)
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duac Low-dose (LD) Gel (N=327) | Clindamycin Gel (N=328) | BPO Gel (N=328) | Vehicle Gel (N=332)
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Ear Congestion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Keratoconus (Eye disorders) | 0 | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dental Caries (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Stomach Discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Application Site Dermatitis (General disorders) | 2 | 0 | 0 | 0
Application Site Dryness (General disorders) | 0 | 0 | 1 | 1
Application Site Eczema (General disorders) | 0 | 0 | 1 | 0
Application Site Erythema (General disorders) | 0 | 0 | 1 | 0
Application Site Hypersensitivity (General disorders) | 0 | 0 | 1 | 0
Application Site Irritation (General disorders) | 1 | 0 | 2 | 0
Application Site Pain (General disorders) | 0 | 1 | 0 | 0
Application Site Photosensitivity Reaction (General disorders) | 2 | 1 | 1 | 2
Application Site Pruritus (General disorders) | 0 | 1 | 1 | 1
Application Site Rash (General disorders) | 0 | 0 | 1 | 0
Drug Intolerance (General disorders) | 0 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0 | 1
Mass (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 2
Hepatic Cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Seasonal Allergy (Immune system disorders) | 0 | 0 | 2 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1
Alveolar Osteitis (Infections and infestations) | 1 | 0 | 0 | 0
Arthritis Infective (Infections and infestations) | 0 | 1 | 0 | 0
Body Tinea (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis Infective (Infections and infestations) | 0 | 0 | 0 | 1
Ear Infection (Infections and infestations) | 1 | 0 | 2 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Fungal Infection (Infections and infestations) | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1 | 2
Gastrointestinal Infection (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Gingival Infection (Infections and infestations) | 0 | 1 | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0
Infectious Mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 3 | 5 | 1 | 4
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 27 | 23 | 32 | 19
Oral Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis Externa (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 2 | 0
Pharyngitis Streptococcal (Infections and infestations) | 0 | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 2 | 2 | 2
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0 | 0
Tinea Infection (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Tooth Abscess (Infections and infestations) | 1 | 0 | 0 | 1
Tooth Infection (Infections and infestations) | 1 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 11 | 13 | 13 | 13
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 1 | 2
Vaginal Infection (Infections and infestations) | 0 | 1 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 1 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1
Fractured Coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 2 | 5 | 0
Limb Crushing Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Neck Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 2
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1
Sunburn (Injury, poisoning and procedural complications) | 2 | 5 | 1 | 2
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood Testosterone Increased (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 8 | 9 | 7
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Sinus Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0
Nephrolithiasis (Psychiatric disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Adnexa Uteri Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Breast Cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1 | 2
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 2
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Chloasma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Elective Surgery (Surgical and medical procedures) | 0 | 0 | 1 | 0
Mole Excision (Surgical and medical procedures) | 1 | 0 | 0 | 0
Tooth Extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1
Wisdom Teeth Removal (Surgical and medical procedures) | 1 | 0 | 2 | 2
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.